CLINICAL TRIAL: NCT04265053
Title: Human Cerebral Blood Flow Regulation: Sex, Mechanism, and Stress Differences
Brief Title: Human Cerebral Blood Flow Regulation
Acronym: Gas Challenge
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-0336; 1R01HL150361-01 (NIH); 21-TRISH PD21-0012 (Other Grant/Funding Number: NASA, HEADQUARTERS (HQ)); A176000 (Other: University of Wisconsin, Madison); EDUC/KINESIOLOGY/KINESIOLOG (Other: University of Wisconsin, Madison); Protocol Version 1, 06/05/2024 (Other: UW Madison)
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-08

CONDITIONS: Cerebral Arterial Diseases
MeSH Terms: conditions — Cerebral Arterial Diseases | interventions — Indomethacin; ganirelix; Estradiol; Antacids

STUDY DESIGN:
Intervention Model Description: Aims 1-2: Both male (n=30) and female (n=27) groups. Participants complete both aims in 2 visits. Participants assigned to one of 2 drug treatments in Aim 2 (n=24/sex/drug). These drugs are mechanistic studies, not treatment studies. Drugs inhibit NOS or COX signaling in blood vessels and are given intravenously during one MRI visit.
  Aim 3: Both male (n=20) and female (n=20) groups (a subset of participants enrolled in Aims 1-2) enroll for ~14 days. All 14 days participants suppress endogenous sex hormones with a GnRH agonist/antagonist, and repeat Aim 1-2 visits around days 5-7. Subsequently, males start taking exogenous testosterone, and females take exogenous estrogen for the remaining 7-9 days. On days 12-14 (depending on MRI and participant schedule), participants repeat visits like Aim 1-2. During half those MRI visits, participants will receive one of the two FDA drugs (same as in original Aim 1-2 visit).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Male NOS (Experimental): Males visit MRI twice. Once for indomethacin visit (hypoxia + hypercapnia), and once for placebo visit (hypoxia + hypercapnia). These 2 MRI visits are conducted in a double-blind placebo controlled design. CBF measured via MRI sequences, and hemodynamics monitored for safety/research.
  Interventions: Drug: Indomethacin 25 MG/50 MG; Drug: Ganirelix Acetate; Drug: Testosterone Transdermal Product; Drug: Antacid
- Male COX (Experimental): Males visit MRI twice. Once for indomethacin visit (hypoxia + hypercapnia), and once for placebo visit (hypoxia + hypercapnia). These 2 MRI visits are conducted in a double-blind placebo controlled design. CBF measured via MRI sequences, and hemodynamics monitored for safety/research.
  Interventions: Drug: Placebo - Lactose; Drug: Ganirelix Acetate; Drug: Testosterone Transdermal Product; Drug: Antacid
- Female NOS (Experimental): Females visit MRI twice. Once for indomethacin visit (hypoxia + hypercapnia), and once for placebo visit (hypoxia + hypercapnia). These 2 MRI visits are conducted in a double-blind placebo controlled design. CBF measured via MRI sequences, and hemodynamics monitored for safety/research.
  Interventions: Drug: Indomethacin 25 MG/50 MG; Drug: Ganirelix Acetate; Drug: Estradiol Topical; Drug: Antacid
- Female COX (Experimental): Females visit MRI twice. Once for indomethacin visit (hypoxia + hypercapnia), and once for placebo visit (hypoxia + hypercapnia). These 2 MRI visits are conducted in a double-blind placebo controlled design. CBF measured via MRI sequences, and hemodynamics monitored for safety/research.
  Interventions: Drug: Placebo - Lactose; Drug: Ganirelix Acetate; Drug: Estradiol Topical; Drug: Antacid

INTERVENTIONS:
Drug: Indomethacin 25 MG/50 MG — Indomethacin is a nonsteroidal anti-inflammatory drug commonly used to reduce fever, pain, stiffness, and swelling from inflammation. It prevents the production of prostaglandins, endogenous signaling molecules known to cause symptoms from inflammation. Indomethacin is used to test COX as a potential mechanism explaining sex differences in CBF control. Indomethacin usage is IND exempt.
  Arms: Female NOS; Male NOS
Drug: Placebo - Lactose — Participants will be screened for lactose intolerance. Total dosing will be calculated to match the mg needed for the indomethacin study visit. Placebo usage is IND exempt.
  Arms: Female COX; Male COX
Drug: Ganirelix Acetate — Gonadotropin-Releasing Hormone (GnRH) antagonist ganirelix acetate as a model to isolate estrogen and testosterone effects on the cerebrovascular system. Participants receive daily injections of ganirelix for 12-14 days for Aim 3 studies only. This will be overseen by clinical endocrinologists.
  Both males and females receive this treatment in Aim 3.
Drug: Testosterone Transdermal Product — In Aim 3, males receive this for 7-9 days of the ganirelix treatment.
  Arms: Male COX; Male NOS
Drug: Estradiol Topical — In Aim 3, females receive this for 7-9 days of the ganirelix treatment.
  Arms: Female COX; Female NOS
Drug: Antacid — Participants will be given a dose of over-the-counter antacid to combat the gastrointestinal distress expected from Indomethacin. Participants will be given a dose of over-the-counter antacid during the placebo visit to mimic the indomethacin study visit. Antacid is IND exempt.

SUMMARY:
This study tests basic differences in how men and women control brain (cerebral) blood flow (CBF), at rest and under stress. The stress is low oxygen or high carbon dioxide. The investigators hypothesize that sex differences per se, plus sex hormone differences, drive different signals in blood vessels that change the way CBF is regulated. The investigators will test these mechanisms with medicine infusions during stress, and measure CBF using state-of-the-art MRI approaches. Research confounding variables like aging and disease will be mitigated by comparing younger adults (18-40 years old).

DETAILED DESCRIPTION:
Cerebrovascular disease is the third leading killer in the U.S., and contributes to decreased quality of life and increased long-term care spending. The risk of cerebrovascular disease is inversely associated with resting cerebral blood flow (CBF). Men exhibit a lower resting CBF and have twice the risk of cerebrovascular disease when compared to premenopausal women. The ability of cerebral vessels to respond to challenges is also inversely related to disease risk, and may be useful in identifying at-risk patients pre-clinically. However, these studies are often confounded by aging and/or comorbidities, and the associations provide little insight into physiologic mechanisms responsible for sexually dimorphic cerebrovascular disease risk. Conversely, animal studies use supraphysiologic levels of hormone treatment in primarily young animals, which limits the translational relevance of animal CBF mechanisms. While there is general agreement that estrogen is protective in healthy adults, the basic impact of sex, and physiologic fluctuations in sex hormones, on mechanisms of CBF control remains unclear.

The overall goal of this research program is to investigate the mechanisms which actively control cerebral blood flow (CBF) in humans, particularly how men and women differ in control mechanisms on a regional basis throughout the brain circulation. The investigators propose to study CBF control mechanisms in healthy younger (18-40 yrs) adult men and women. The overall hypothesis is that female sex and sex hormones contribute to larger stress-induced increases in CBF, due to greater prostanoid (COX) and nitric oxide (NOS) dilation.

A key technological innovation of this proposal derives from multi-mode, high-resolution, flow sensitive MRI to quantify CBF at macrovascular and microvascular levels, at rest, and in response to environmental challenges (stress test for the brain). Additionally, the research design allows for quantification of sex differences in two vascular control mechanisms across all brain regions. Preliminary data demonstrate: hypoxic cerebral vasodilation is 60-100% higher in women compared to men, COX inhibition reduces dilation in women but not men, NOS inhibition reduces vasodilation more in women. Those concepts will be tested in Aims 1-2 of the grant in this current proposal, covered in Phase 1 using technical innovative MRI and pharmacologic tools to test potential sex specific mechanisms of CBF control. The conceptual innovation is planned in Aim 3 of the grant (or Phase 2). Participants must complete Phase 1 studies to continue to Phase 2. Study procedures in Phase 1 and 2 are identical, but the investigators conduct them twice: once in the context of sex hormone suppression, and a second time during a single hormone replacement (during suppression), to study the independent impact of testosterone (men) and estrogen (women) on CBF control mechanisms.

Substantial preliminary findings support these hypotheses, and integrated physiologic, pharmacologic, and MRI approaches are available to test them. This state-of-the-art approach will yield previously unattainable insight into not only maintaining basal CBF, but actively controlling it during physiologic demands for increased flow. These novel, high resolution, regionally-specific, sex-specific, and mechanism-specific findings will serve as a knowledge platform, for designing sex-specific CBF studies in high risk disease populations (e.g. diabetes, hypertension, Alzheimer's) which exhibit strong sex-specific etiology and important vascular contributions. To assess the effects of sex hormones on the microbiome, the investigators will also be collecting fecal samples from participants before hormone manipulation, after hormone suppression, and after single hormone add-back.

Three Specific Aims will be addressed in this study:

Aim 1: Test the hypothesis that healthy males exhibit reduced cerebral vasodilation compared to healthy females despite exhibiting similar vasodilation to hypercapnia.

* Aim 1A: Vasodilation to hypoxia will be markedly lower in males, more so in anterior brain regions.
* Aim 1B: Vasodilation to hypercapnia will be similar between sexes.

Aim 2: Test the hypothesis that acute inhibition of COX or NOS will reduce sex differences in hypoxia-mediated cerebral vasodilation.

* Aim 2A: COX-mediates vasodilation primarily in females.
* Aim 2B: NOS mediates vasodilation more in females than males.

Aim 3: Test the hypothesis that manipulating sex steroids can abolish or magnify sex differences in vasodilation.

* Aim 3A: Short-term suppression of sex steroids will abolish sex differences in resting and hypoxic CBF via greater losses of COX- and NOS-mediated vasodilation in females than males.
* Aim 3B: Short-term supplementation of unopposed testosterone in males will magnify sex differences by driving COX vasoconstriction (TXA2) and uncoupled NOS vasoconstriction.
* Aim 3C: Short-term supplementation of unopposed estradiol in females will magnify sex differences via increased NOS and COX vasodilation.

Updated Protocol (CP011):

Fifty-four (54) otherwise healthy adults between 18-40 years of age inclusive composed of 27 males and 27 females. These 54 participants will complete both Aims 1 and 2 (both Aims completed in 2 study visits).

Updated Protocol (CP017):

Fifty-seven (57) otherwise healthy adults between 18-40 years of age inclusive composed of 30 males and 27 females. These 57 participants will complete both Aims 1 and 2 (both Aims completed in 2 study visits). The number of male participants was increased by 3 to meet the recruitment requirements of the Phase 2 (2023-0548) study. Completion of Phase 1 (2020-0336) is required to participate in Phase 2. No females were added as the recruitment for Phase 2 females will fall within the 27 females who will have completed Phase 1 (2020-0336).

ELIGIBILITY:
Inclusion Criteria:

* All participants will be healthy adults between 18-40 years old, matched for age and aerobic fitness
* Participants will be non-hypertensive (<125/80mm Hg)
* Participants will be non-obese (BMI 19-25 kg/m2)
* Participants will have normal blood glucose (<100 g/dl)
* Participants will have normal lipids (LDL cholesterol <130 mg/dl, triglycerides <150 mg/dl)
* Women must have a natural regular menstrual cycle

Exclusion Criteria:

* Participants with a history of:

  * peripheral vascular disease
  * hepatic disease
  * renal disease
  * hematologic disease
  * stroke
  * obesity
  * prediabetes
  * diabetes
  * sleep apnea
* Participants with current BP>130/85 mmHg
* Regular smokers
* Taking cardiovascular medications
* Women who take hormonal birth control
* Women who are pregnant or have polycystic ovarian syndrome [Hormonal birth control will not be allowed in women]
* Contradictions to MRI
* Lactose intolerance

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Cerebrovascular Conductance (CVC) in response to Hypoxia | up to 75 minutes for entire visit, but hypoxia lasts about 20 minutes
  CVC is the ratio between Cerebral Blood Flow (CBF) and blood pressure (BP). Change in CVC in response to hypoxia between male and female groups, where baseline CVC is subtracted from hypoxia CVC. Hypoxia typically lasts about 20 minutes. The hypothesis is that women will exhibit 50-60% more vasodilation in response to hypoxia [Aim 1].
CVC in response to Hypercapnia | up to 75 minutes for entire visit, but hypercapnia lasts about 10-15 minutes
  CVC is the ratio between Cerebral Blood Flow (CBF) and blood pressure (BP). Change in CVC in response to hypercapnia between male and female groups, where CBF is normalized for BP. Baseline CVC will be subtracted from hypercapnia CVC. Hypercapnia typically lasts about 10-15 minutes.The hypothesis is that hypercapnic vasodilation will be similar between groups [Aim 1B].
CVC change in response to Drug Infusion | approximately 10 minutes in the middle of 75 minute study visit
  CVC is the ratio between Cerebral Blood Flow (CBF) and blood pressure (BP). Change in CVC in response to drug infusion between male [NOS or COX] and female [NOS or COX] groups. The hypothesis is that acute inhibition of COX or NOS will reduce sex differences in hypoxia-mediated cerebral vasodilation [Aim 2].
Change in hypoxia CVC in response to Ganirelix compared to no ganirelix Baseline (Aim 3a) | baseline and up to 7 days during ganirelix treatment
  Change in hypoxia CVC response to ganirelix compared to baseline within male and female groups, where CVC is CBF is normalized for BP. The hypothesis is that GnRH suppression will abolish hypoxic CBF differences, indicating sex steroids play a vital role in CBF control [Aim 3].
Change in hypoxia CVC response to sex hormone suppression with single sex hormone add-back | baseline and up to 14 days
  Change in hypoxia CVC response to ganirelix+testosterone (in males Aim 3B) or ganirelix+estradiol (in females, Aim 3C) compared to baseline within male and female groups, where CVC is CBF is normalized for BP. The hypothesis is that adding a sex steroid will magnify hypoxic CVC differences, indicating sex steroids play a vital role in CBF control [Aim 3].
Change in hypoxia CVC response to NOS or COX inhibition during ganirelix+single sex hormone add-back | baseline and up to 14 days
  Change in hypoxia CVC drug response to NOS or COX inhibition during ganirelix+testosterone (in males Aim 3B) or ganirelix+estradiol (in females, Aim 3C) compared to baseline hypoxia studies from Aim 2. The hypothesis is that adding a sex steroid will magnify hypoxic CVC differences in drug effects, indicating sex steroids play a vital role in CBF control [Aim 3].

CONTACTS AND LOCATIONS:
Overall Officials: William Schrage, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No